CLINICAL TRIAL: NCT03123107
Title: Advancing the Cardiovascular Science of Vitamin C in Cardiac Surgery Patients
Brief Title: Vitamin C in Cardiac Surgery Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Wilkes University (Other)
Responsible Party: Principal Investigator, Deepak Singh, Principal Investigator, Geisinger Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-0463
Record Dates: First submitted 2017-04-05; First posted 2017-04-21 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: Vitamin C; Postoperative atrial fibrillation; coronary artery bypass graft; ascorbic acid
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ascorbic Acid (Experimental): 4 patients will receive 15 mg/kg of ascorbic acid IV the day before and after CABG surgery; 4 patients will receive 30 mg/kg of ascorbic acid IV the day before and after CABG surgery. The maximum dose of ascorbic acid will be 2 g.
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic acid doses will be mixed in 100 mL normal saline and infused over 60 minutes. The postoperative dose will be given on postoperative day #1.
  Other Names: Vitamin C

SUMMARY:
Postoperative atrial fibrillation (POAF) is a common complication following cardiac surgery that increases the incidence of stroke, kidney injury and death. Vitamin C has been shown to decrease the incidence of POAF follow cardiac surgery, but the optimal dose has not been identified. With this project, the investigators plan to gather pharmacokinetic and dose-response data for vitamin C in the cardiac surgery population. The investigators plan to conduct a small interventional pilot study investigating the pharmacokinetics and pharmacodynamics of Vitamin C in patients undergoing coronary artery bypass graft (CABG) surgery. Patients enrolled will receive an intravenous dose of Vitamin C the day before surgery and the day after. Patients will have blood samples obtained with each dose for analysis of vitamin C concentrations and several biomarkers of oxidative stress. Analysis of samples will be performed within the Department of Pharmaceutical Sciences at Wilkes University.

DETAILED DESCRIPTION:
The pathophysiology of post-operative atrial fibrillation (POAF) in cardiac surgery patients has not been fully elucidated, but inflammation and oxidative stress are associated with its occurrence. Increased activity of nicotinamide adenine dinucleotide phosphate (NADPH) oxidase and production of glutathione and nitrotyrosine have been found to occur in animal models of atrial fibrillation and patients who develop POAF. Similarly, malondialdehyde (MDA), a biomarker of lipid peroxidation, has also been shown to increase during cardiac surgery, and be significantly more elevated in patients who develop POAF. Cardiac surgery patients supplemented with ascorbic acid have reduced expression of NADPH oxidase and levels of MDA, glutathione and nitrotyrosine, and reduced POAF rates. Ascorbic acid supplementation has demonstrated a significant reduction in POAF in small clinical trials enrolling patients undergoing cardiac surgery. Collectively, these findings show that ascorbic acid prevents POAF in a novel way compared to recommended therapies such as beta-blockers and amiodarone, without the risk of significant side effects. However, the doses of ascorbic acid utilized in clinical trials have been found to inadequately suppress the production of inflammatory markers associated with POAF. Therefore, the maximum effect of ascorbic acid for POAF prevention may not have been realized in clinical trials published to date. These suboptimal responses may be attributable to known variances in medication pharmacokinetics in the cardiac surgery population that lead to reduced medication bioavailability, metabolism and elimination. The variation in ascorbic acid pharmacokinetics in this population is unknown. Thus, the contribution of the proposed research is expected to be determination of the pharmacokinetic profile of ascorbic acid and its concentration-response relationship with oxidative biomarkers associated with POAF in the cardiac surgery population.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21 to 79 years of age admitted to Geisinger Wyoming Valley (GWV) and scheduled to undergo urgent CABG
* Planned utilization of cardiopulmonary bypass during the surgical procedure

Exclusion Criteria:

* Body mass index greater than 30 kg/m2
* Estimated creatinine clearance less than 30 ml/min
* History of persistent or permanent atrial fibrillation
* Condition associated with oxidative stress or inflammation (e.g. chronic rheumatic, inflammatory or neoplastic disease, recent infection, etc.)
* Currently taking corticosteroids, non-steroidal anti-inflammatory drugs or deferoxamine
* History of oxalate kidney stones
* Currently pregnant
* History of allergic reaction to ascorbic acid products
* Currently taking any herbals or supplements (not including a multivitamin or calcium)
* Enrolled in another research study

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Ascorbate maximum serum concentration (Cmax) | 1 year
  Maximum serum concentration of ascorbate obtained after drug administration.
Half-life of serum ascorbate (T1/2) | 1 year
  The amount of time is takes for the serum concentration of ascorbate to decrease by half.
Elimination rate constant of ascorbate (Ke) | 1 year
  The rate at which ascorbate is eliminated from the body
Area under the concentration-time curve for serum ascorbate (AUC) | 1 year
  Describes the overall concentration in the body given an administered dose of ascorbic acid.
Change in biomarker concentrations | Change within 24 hours; preoperative compared to postoperative
  This will consist of the concentrations of NADP+, NADPH, MDA, GGS and nitrotyrosine in blood and atrial tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Singh, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoniades C, Demosthenous M, Reilly S, Margaritis M, Zhang MH, Antonopoulos A, Marinou K, Nahar K, Jayaram R, Tousoulis D, Bakogiannis C, Sayeed R, Triantafyllou C, Koumallos N, Psarros C, Miliou A, Stefanadis C, Channon KM, Casadei B. Myocardial redox state predicts in-hospital clinical outcome after cardiac surgery effects of short-term pre-operative statin treatment. J Am Coll Cardiol. 2012 Jan 3;59(1):60-70. doi: 10.1016/j.jacc.2011.08.062. PMID 22192670
- [Background] Bruins P, te Velthuis H, Yazdanbakhsh AP, Jansen PG, van Hardevelt FW, de Beaumont EM, Wildevuur CR, Eijsman L, Trouwborst A, Hack CE. Activation of the complement system during and after cardiopulmonary bypass surgery: postsurgery activation involves C-reactive protein and is associated with postoperative arrhythmia. Circulation. 1997 Nov 18;96(10):3542-8. doi: 10.1161/01.cir.96.10.3542. PMID 9396453
- [Background] Carnes CA, Chung MK, Nakayama T, Nakayama H, Baliga RS, Piao S, Kanderian A, Pavia S, Hamlin RL, McCarthy PM, Bauer JA, Van Wagoner DR. Ascorbate attenuates atrial pacing-induced peroxynitrite formation and electrical remodeling and decreases the incidence of postoperative atrial fibrillation. Circ Res. 2001 Sep 14;89(6):E32-8. doi: 10.1161/hh1801.097644. PMID 11557745
- [Background] Castillo R, Rodrigo R, Perez F, Cereceda M, Asenjo R, Zamorano J, Navarrete R, Villalabeitia E, Sanz J, Baeza C, Aguayo R. Antioxidant therapy reduces oxidative and inflammatory tissue damage in patients subjected to cardiac surgery with extracorporeal circulation. Basic Clin Pharmacol Toxicol. 2011 Apr;108(4):256-62. doi: 10.1111/j.1742-7843.2010.00651.x. Epub 2010 Dec 8. PMID 21138533
- [Background] Colby JA, Chen WT, Baker WL, Coleman CI, Reinhart K, Kluger J, White CM. Effect of ascorbic acid on inflammatory markers after cardiothoracic surgery. Am J Health Syst Pharm. 2011 Sep 1;68(17):1632-9. doi: 10.2146/ajhp100703. PMID 21856809
- [Background] Dehghani MR, Majidi N, Rahmani A, Asgari B, Rezaei Y. Effect of oral vitamin C on atrial fibrillation development after isolated coronary artery bypass grafting surgery: A prospective randomized clinical trial. Cardiol J. 2014;21(5):492-9. doi: 10.5603/CJ.a2013.0154. Epub 2013 Dec 2. PMID 24293167
- [Background] Dingchao H, Zhiduan Q, Liye H, Xiaodong F. The protective effects of high-dose ascorbic acid on myocardium against reperfusion injury during and after cardiopulmonary bypass. Thorac Cardiovasc Surg. 1994 Oct;42(5):276-8. doi: 10.1055/s-2007-1016504. PMID 7863489
- [Background] Dudley SC Jr, Hoch NE, McCann LA, Honeycutt C, Diamandopoulos L, Fukai T, Harrison DG, Dikalov SI, Langberg J. Atrial fibrillation increases production of superoxide by the left atrium and left atrial appendage: role of the NADPH and xanthine oxidases. Circulation. 2005 Aug 30;112(9):1266-73. doi: 10.1161/CIRCULATIONAHA.105.538108. PMID 16129811
- [Background] Eslami M, Badkoubeh RS, Mousavi M, Radmehr H, Salehi M, Tavakoli N, Avadi MR. Oral ascorbic acid in combination with beta-blockers is more effective than beta-blockers alone in the prevention of atrial fibrillation after coronary artery bypass grafting. Tex Heart Inst J. 2007;34(3):268-74. PMID 17948074
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Kim YM, Guzik TJ, Zhang YH, Zhang MH, Kattach H, Ratnatunga C, Pillai R, Channon KM, Casadei B. A myocardial Nox2 containing NAD(P)H oxidase contributes to oxidative stress in human atrial fibrillation. Circ Res. 2005 Sep 30;97(7):629-36. doi: 10.1161/01.RES.0000183735.09871.61. Epub 2005 Aug 25. PMID 16123335
- [Background] Kim YM, Kattach H, Ratnatunga C, Pillai R, Channon KM, Casadei B. Association of atrial nicotinamide adenine dinucleotide phosphate oxidase activity with the development of atrial fibrillation after cardiac surgery. J Am Coll Cardiol. 2008 Jan 1;51(1):68-74. doi: 10.1016/j.jacc.2007.07.085. PMID 18174039
- [Background] Mihm MJ, Yu F, Carnes CA, Reiser PJ, McCarthy PM, Van Wagoner DR, Bauer JA. Impaired myofibrillar energetics and oxidative injury during human atrial fibrillation. Circulation. 2001 Jul 10;104(2):174-80. doi: 10.1161/01.cir.104.2.174. PMID 11447082
- [Background] Papoulidis P, Ananiadou O, Chalvatzoulis E, Ampatzidou F, Koutsogiannidis C, Karaiskos T, Madesis A, Drossos G. The role of ascorbic acid in the prevention of atrial fibrillation after elective on-pump myocardial revascularization surgery: a single-center experience--a pilot study. Interact Cardiovasc Thorac Surg. 2011 Feb;12(2):121-4. doi: 10.1510/icvts.2010.240473. Epub 2010 Nov 23. PMID 21098510
- [Background] Pea F, Pavan F, Furlanut M. Clinical relevance of pharmacokinetics and pharmacodynamics in cardiac critical care patients. Clin Pharmacokinet. 2008;47(7):449-62. doi: 10.2165/00003088-200847070-00002. PMID 18563954
- [Background] Ramlawi B, Otu H, Mieno S, Boodhwani M, Sodha NR, Clements RT, Bianchi C, Sellke FW. Oxidative stress and atrial fibrillation after cardiac surgery: a case-control study. Ann Thorac Surg. 2007 Oct;84(4):1166-72; discussion 1172-3. doi: 10.1016/j.athoracsur.2007.04.126. PMID 17888965
- [Background] Rodrigo R, Korantzopoulos P, Cereceda M, Asenjo R, Zamorano J, Villalabeitia E, Baeza C, Aguayo R, Castillo R, Carrasco R, Gormaz JG. A randomized controlled trial to prevent post-operative atrial fibrillation by antioxidant reinforcement. J Am Coll Cardiol. 2013 Oct 15;62(16):1457-65. doi: 10.1016/j.jacc.2013.07.014. Epub 2013 Jul 31. PMID 23916928